CLINICAL TRIAL: NCT02376946
Title: Evaluation of Postoperative Edema and Pain Following Third Molar Extraction With Application of Pulsed Electromagnetic Field (PEMF) Therapy
Brief Title: Third Molar Extraction and Pulsed Electromagnetic FieldTherapy
Acronym: PEMF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Tufts University (Other)
Collaborators: BioElectronics Corporation (Industry)
Responsible Party: Principal Investigator, Archana Viswanath, Assistant Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 10436
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Edema and Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Actipatch (Active Comparator): The study group will be comprised of subjects that will receive PEMF ActiPatchTM treatment for postoperative management of pain and edema.
  Interventions: Device: ActiPatch(TM)
- Placebo (Placebo Comparator): The control group will be comprised of the subjects that will receive a placebo patch as treatment for postoperative management of pain and edema.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: ActiPatch(TM) — Assigned by randomization, this study group will be comprised of subjects that receive the PEMF ActiPatch(TM) treatment for postoperative management of pain and edema.
  Other Names: ActiBand(TM)
  Arms: Actipatch
Device: Placebo — Assigned by randomization, this control group will be comprised of the subjects that receive a placebo patch as treatment for postoperative management of pain and edema.
  Arms: Placebo

SUMMARY:
This study is a prospective, randomized, double-blinded, controlled, clinical trial that evaluates the efficacy of using PEMF in the postoperative period in decreasing swelling and pain after extraction of impacted third molars. The study group will be comprised of subjects that will receive PEMF Actiband treatment for postoperative management of pain and edema. The control group will be comprised of the subjects that will receive a placebo patch as treatment for postoperative management of pain and edema.

Thirty (30) subjects will be randomly assigned to each group. Enrollment will continue until 60 qualified subjects have been recruited. Eligibility criteria will be based on the standards for conducting oral surgery procedures on third molar extractions, in addition to safety considerations and contraindications for the Actiband and other agents to be used. Moreover, the selected subjects will have the same surgical difficulty and surgical trauma anticipated standardized by classification system of impacted third molars. All inclusion and exclusion criteria will be thoroughly explained in the relevant section of this proposal. Postoperative edema and pain will be evaluated using 3dMD and Visual Analog Scale, respectively. Different measurements will be obtained immediately before the surgery and in standard periodic intervals as described in the Materials and Methods section of the proposal. Any difference in postoperative edema, pain, and site responsible for request of rescue pain medication will be compared and analyzed between the two groups.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blinded, controlled, clinical trial that evaluates the efficacy of using PEMF in the postoperative period in decreasing swelling and pain after extraction of partial or full/complete boney impacted third molars. The study group will be comprised of subjects that will receive PEMF ActiPatchTM treatment for postoperative management of pain and edema. The control group will be comprised of the subjects that will receive a placebo patch as treatment for postoperative management of pain and edema.

Thirty (30) subjects will be randomly assigned to each group. Enrollment will continue until sixty (60) qualified subjects have been recruited. Eligibility criteria will be based on the standards for conducting oral surgery procedures on third molar extractions, in addition to safety considerations and contraindications for the ActiPatch(TM) and other agents to be used. Moreover, the selected subjects will have the same surgical difficulty and surgical trauma anticipated standardized by classification system of impacted third molars. This classification system is utilized in the TUSDM (Tufts University School of Dental Medicine) oral surgery clinic. All inclusion and exclusion criteria will be thoroughly explained in the relevant section of this proposal. Postoperative edema and pain will be evaluated using 3dMD(TM) and Visual Analog Scale, respectively. Different measurements will be obtained immediately before the surgery and in standard periodic intervals as described in the Materials and Methods section of the proposal. Any difference in postoperative edema, pain, and site responsible for request of rescue pain medication will be compared and analyzed between the two groups.

Up to 200 subjects will be enrolled in the study to account for screen failures. Up to forty (40) subjects will be randomly assigned to each group. Recruitment will continue until up to eighty (80) subjects have qualified for study participation. This will allow for up to 25% dropout to end with 60 subjects completing the study.

The primary outcome, postoperative facial swelling at 72 hours (as measured by the 3dMD(TM)), will be compared between the two groups using independent sample t-test if the data are normally distributed, or the Mann Whitney U test if non-parametric methods need to be utilized. This approach will also be utilized for comparing pain (as measured by VAS). The percentage of subjects who will use rescue pain medication due to experience of postoperative pain on the group treated with PEMF ActiPatch(TM) will be compared with the percentage of subjects who will use rescue pain medication due to experience of postoperative pain for the group received placebo, using a Chi-square test. In addition, the volume measurements and the VAS scores will be analyzed using a repeated measures analysis, adjusting for subject age, gender and pain perception. Furthermore, a correlation between placebo group and the use of rescue pain medication will be determined and the association will be dictated by calculating the odds ratio. The statistical significance of this association will be examined using the Chi-square test. All p-values less than 0.025 will be considered statistically significant. Statistical analyses will be performed using SAS, Version 9.2 (SAS Institute, Cary, NC).

An initial 3dMD(TM) scan will be obtained for baseline evaluation at the extraction visit. A second 3dMD(TM) scan will be obtained for evaluation and determination of facial swelling at the 72 hour follow up visit. A third scan will be obtained at the 10 day follow up visit to evaluate the degree of resolution of swelling. The scan will result in a computer-generated image, on which the investigator will outline the area of clinical interest and calculate the volume using integration. The process of surface scanning and volume measurement will use the 3dMD(TM) Vultus software® (3dMD(TM), Atlanta, Georgia, United States).The Vultus software allows for pre and post-surgery superimposition of images as well as quantitative evaluation of surface and volume changes. The PI has had on site training at the Georgia 3dMD facility and had additional training when the camera array was installed. The technique of obtaining the image is straight forward and there is a set of instructions at the installation site for immediate review as necessary. The PI and a representative from 3dMD company will give training to the co-investigators who will be using the device.

The degree of facial swelling between the two groups at the two time points (72 hour follow up and 10 day follow up) will be compared using the data collected from 3dMD(TM). Furthermore, the change in volume between the two scans taken at the 72 hour follow up visit and the 10 day follow up within each group will also be compared. The volumetric difference between the two groups will be analyzed for any statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex and of any race between the ages of 18 and 30 years. 30 Years old is the upper age limit because wisdom teeth extraction is normally done between the ages of 18 and 30, since after the age of 30 additional complications can arise during surgeries.
2. Subjects for whom a decision has been made to extract 2 to 4 third molars. At least two must be classified as full or partially bony impacted (as defined below) of any angulation under local anesthesia alone, local anesthesia and sedation or local anesthesia and general anesthesia all in an outpatient setting.

   1. Full/complete bony: The entire tooth is below the level of the alveolar bone. The tooth is completely encased in bone so that when the gingiva is cut and reflected back, the tooth is not seen. Bone removal (large amounts) together with root sectioning will be needed to remove the tooth.33
   2. Partial bony: A portion of the height of the contour of the tooth is below the level of the alveolar bone. The superficial portion of the tooth is covered only by soft tissue but the height of the tooth's contour is below the level of the surrounding alveolar bone.33
3. Subjects must be physically able to tolerate conventional surgical procedures (ASA I/II)
4. Subjects must agree to follow the study protocol.

Exclusion Criteria:

1. Subjects who are known to be pregnant or think they may be pregnant. (A urine pregnancy test will be performed on female subjects at Day 0 - Visit 1. Subjects testing positive will be excluded from study participation.
2. Subjects with a cardiac pacemaker, cardioverter defibrillator, neurostimulator or any active medical or metallic implant (including dental implant).
3. Subjects with skeletal immaturity.
4. Subjects with self-reported current or history of substance abuse.
5. Subjects who are currently receiving any anti-inflammatory or pain medication chronically or they suffer from a chronic pain condition.
6. Subjects with an allergy to vicodin (or its constituents, acetaminophen and hydrocodone).
7. Subjects who are diagnosed with fibromyalgia.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Archana Viswanath, Principal Investigator — Research Professor
Locations (1):
- Tufts University School of Dental Medicine Department of Oral and Maxillofacial Surgery, Boston, Massachusetts, United States

REFERENCES:
- [Background] Little RC, Ginsburg JM. The physiologic basis for clinical edema. Arch Intern Med. 1984 Aug;144(8):1661-4. doi: 10.1001/archinte.144.8.1661. PMID 6466021
- [Background] Conrad SM, Blakey GH, Shugars DA, Marciani RD, Phillips C, White RP Jr. Patients' perception of recovery after third molar surgery. J Oral Maxillofac Surg. 1999 Nov;57(11):1288-94; discussion 1295-6. doi: 10.1016/s0278-2391(99)90861-3. PMID 10555792
- [Background] van Gool AV, Ten Bosch JJ, Boering G. Clinical consequences of complaints and complications after removal of the mandibular third molar. Int J Oral Surg. 1977 Feb;6(1):29-37. doi: 10.1016/s0300-9785(77)80069-0. PMID 402320
- [Background] Zuniga JR, Phillips CL, Shugars D, Lyon JA, Peroutka SJ, Swarbrick J, Bon C. Analgesic safety and efficacy of diclofenac sodium softgels on postoperative third molar extraction pain. J Oral Maxillofac Surg. 2004 Jul;62(7):806-15. doi: 10.1016/j.joms.2003.12.019. PMID 15218558
- [Background] Urquhart E. Analgesic agents and strategies in the dental pain model. J Dent. 1994 Dec;22(6):336-41. doi: 10.1016/0300-5712(94)90084-1. PMID 7844260
- [Background] Mehlisch DR. The efficacy of combination analgesic therapy in relieving dental pain. J Am Dent Assoc. 2002 Jul;133(7):861-71. doi: 10.14219/jada.archive.2002.0300. PMID 12148679
- [Background] Troullos ES, Hargreaves KM, Butler DP, Dionne RA. Comparison of nonsteroidal anti-inflammatory drugs, ibuprofen and flurbiprofen, with methylprednisolone and placebo for acute pain, swelling, and trismus. J Oral Maxillofac Surg. 1990 Sep;48(9):945-52. doi: 10.1016/0278-2391(90)90007-o. PMID 2395047
- [Background] Schultze-Mosgau S, Schmelzeisen R, Frolich JC, Schmele H. Use of ibuprofen and methylprednisolone for the prevention of pain and swelling after removal of impacted third molars. J Oral Maxillofac Surg. 1995 Jan;53(1):2-7; discussion 7-8. doi: 10.1016/0278-2391(95)90486-7. PMID 7799116
- [Background] Ganzber S. Analgesics: opioids and nonopioids. In: Ciancio S, ed. ADA guide to dental therapeutics. Chicago: ADA Publishing; 1998:80-107.
- [Background] Dionne RA, Gordon SM. Nonsteroidal anti-inflammatory drugs for acute pain control. Dent Clin North Am. 1994 Oct;38(4):645-67. PMID 7805940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Actipatch | Placebo
Started | 0 (study terminated prior to being conducted) | 0 (study terminated prior to being conducted)
Completed | 0 (study terminated prior to being conducted) | 0 (study terminated prior to being conducted)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: study terminated prior to being conducted
Groups:
- Total: Total of all reporting groups
Arm/Group | Actipatch | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Postoperative Facial Swelling
Description: The primary outcome, postoperative facial swelling at 72 hours (as measured by the 3dMDTM), will be compared between the two groups using independent sample t-test if the data are normally distributed, or the Mann Whitney U test if non-parametric methods need to be utilized.
Time Frame: 72 Hours post surgery and 10 days post surgery
Population: study terminated prior to being conducted
Arm/Group | Actipatch | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: study terminated prior to being conducted
Description: study terminated prior to being conducted
Arm/Group | Actipatch | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes